CLINICAL TRIAL: NCT06489210
Title: A Comparison Between Posterior, Lateral and Medial Approaches for Ultrasound-guided Popliteal Block: A Randomized Clinical Study
Brief Title: A Comparison Between Posterior, Lateral and Medial Approaches for Ultrasound-guided Popliteal Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Adel Ali Hassan, lecturer of anaesthesia, intensive care and pain management, Helwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4428-4-3-2018
Record Dates: First submitted 2024-06-20; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Nerve Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- popliteal block posterior approach group (Active Comparator): through posterior approach ultrasound guided sciatic nerve block at popliteal fossa 20ml of the selected local anesthetic mixture (10ml of 0.5% bupivacaine mixed with 10ml of 2% lidocaine, each with 1:200,000 epinephrine) was injected incrementally
  Interventions: Procedure: popliteal block
- popliteal block lateral approach group (Active Comparator): ultrasound guided sciatic nerve block at popliteal fossa through lateral approach 20ml of the selected local anesthetic mixture (10ml of 0.5% bupivacaine mixed with 10ml of 2% lidocaine, each with 1:200,000 epinephrine) was injected incrementally
  Interventions: Procedure: popliteal block
- poplitea block medial approach group (Active Comparator): ultrasound guided sciatic nerve block at popliteal fossa through medial approach 20ml of the selected local anesthetic mixture (10ml of 0.5% bupivacaine mixed with 10ml of 2% lidocaine, each with 1:200,000 epinephrine) was injected incrementally
  Interventions: Procedure: popliteal block

INTERVENTIONS:
Procedure: popliteal block — using ultrasound to detect sciatic nerve and popliteal fossa through different approaches using 20ml of the selected local anesthetic mixture (10ml of 0.5% bupivacaine mixed with 10ml of 2% lidocaine, each with 1:200,000 epinephrine) was injected incrementally

SUMMARY:
Background: Popliteal block is a widely used technique to provide anesthesia or analgesia for below-knee surgical procedures. In this study, the investigators compare ultrasound-guided popliteal blocks via posterior, lateral, and medial approaches to find out the approach with the best outcome.

DETAILED DESCRIPTION:
Methods: In this randomized, controlled clinical trial, one hundred and twenty ASA physical status of class I and II patients undergoing below-knee surgery were involved. These patients were divided into three equal groups at randomly based on the route assigned for the US-guided popliteal block: the posterior, lateral, and medial approach groups. In this study, technical characteristics [number of attempts to get the proper injection site and block performance time], anesthetic and analgesic characteristics [success rate, block onset, potency, and duration, time to ask, and the consumed amount of postoperative analgesia], discomfort rate in respect to position and needle insertion and the associated complications were recorded.

ELIGIBILITY:
Inclusion Criteria: This study included

* ASA physical status (PS) class I and II
* weighing 70-85 kg,
* undergoing elective below knee surgeries

Exclusion Criteria:

* patients who refused to participate in the study
* those having an allergy to local anesthetics
* peripheral neuropathy, coagulopathy
* diabetes mellitus
* severe hepatic
* renal impairment
* infection, mass and crush injury or open wound at the nerve block site
* patients receiving chronic analgesic therapy.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
assessment of intraoperative and postoperative pain in different groups after intervention | 24 hours after operation
  pain severity levels via visual analogue scale (VAS). VAS is a 10 cm horizontal line labeled "no pain" at one end and "worst pain" imaginable on the other end. The patient was asked to mark on this line where the intensity of the patient lies

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University Hospitals, Zagazig, Egypt